CLINICAL TRIAL: NCT02593487
Title: Effect of Rosuvastatin Therapy on HDL2 Level and Antiatherosclerotic Reverse Cholesterol Transport Process in Chinses CAD Patients With Hyperlipidemia
Brief Title: Effect of Rosuvastatin Therapy on HDL2 Level
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Xu-kai Wang, MD，PhD, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ESR-14-10333
Record Dates: First submitted 2015-10-29; First posted 2015-11-02 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-10

CONDITIONS: Hyperlipemia; Coronary Heart Disease
Keywords: Coronary Artery Disease; Hyperlipidemia; Rosuvastatin; Lipoproteins; high-density lipoprotein; HDL2
MeSH Terms: conditions — Hyperlipidemias; Coronary Disease; Coronary Artery Disease | interventions — Rosuvastatin Calcium; Population Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rosuvastatin 10mg/d group (Experimental): rosuvastatin 10mg table by mouth, qd
  Interventions: Drug: Rosuvastatin 10mg/d group
- Rosuvastatin 20mg/d group (Active Comparator): rosuvastatin 20mg table by mouth, qd
  Interventions: Drug: Rosuvastatin 20mg/d group

INTERVENTIONS:
Drug: Rosuvastatin 10mg/d group — rosuvastatin 10mg tablet,q.d. for 12 weeks.
  Other Names: Routine dose group
  Arms: Rosuvastatin 10mg/d group
Drug: Rosuvastatin 20mg/d group — rosuvastatin 20mg tablet,q.d. for 12 weeks.
  Other Names: Loading dose group
  Arms: Rosuvastatin 20mg/d group

SUMMARY:
In many large trials, reducing low density lipoprotein (LDL) levels with rosuvastatin decreased the incidence of major cardiovascular events，but little attention to the effects of rosuvastatin on HDL level，especially on HDL subtype.

Epidemiological evidence strongly favors the notion that the risk of cardiovascular disease (CVD) is inversely related to the plasma high-density lipoprotein (HDL) cholesterol concentration.

HDL can be subdivided into large-sized (HDL2a, HDL2b) and small-sized subclasses (preb1-HDL, HDL3c, HDL3b, HDL3a) and preb2-HDL. Some studies indicate that only large HDL2a and HDL2b particles make HDLs possess anti-atherogenic functions.

The investigators assume that rosuvastatin could play the role of anti-atherosclerosis though the levels of HDL2a、HDL2b increased.

DETAILED DESCRIPTION:
Elevated LDL-C and lowered HDL-C are important risk factors for cardiovascular disease. Raising HDL-C is an attractive approach for reducing the residual risk of cardiovascular events that persist in many patients receiving low-density LDL-C -lowering therapy with statins. From previous studies, it is concluded that compared to atorvastatin, rosuvastatin could significantly increase HDL-C levels from baseline. However, which benefits the elevated HDL-C will bring to these patients who receive statin lowing LDL-C therapy are still unknown. Despite strong evidence that HDL-C levels predict atherosclerotic events, attempts at using an HDL-based treatment strategy as a therapeutic target have not yet been successful at the present time. However, on the basis of an enormous amount of basic scientific and clinical investigation, the International Atherosclerosis Society and US National Lipid Association still believe that there are a considerable number of reasons supporting the need to continue to investigate the therapeutic effect of modulating HDL structure and function.

It has long been known that a low level of HDL cholesterol is a powerful independent predictor of increased cardiovascular risk, even among patients with LDL cholesterol levels below 70 mg/dl. In fact, a 1 mg/dl (0.026 mM) increment in HDL-C levels was associated with a significant decrease in the risk of coronary heart disease (CAD) of 2% in men and 3% in women. HDL-C has been proposed to have several anti-atherosclerotic properties, including the ability to mediate reverse cholesterol transport (RCT), antioxidant capacity, anti-inflammatory properties, nitric oxide-promoting activity, and an ability to transport proteins with their own intrinsic biological activities. RCT describes the metabolism and an important antiatherogenic function of HDL, namely, the HDL-mediated efflux of cholesterol from cells of the arterial wall and its subsequent delivery to the liver and steroidogenic organs, thus preventing atherosclerosis. HDL particles are responsible for RCT, as critical acceptors of cholesterol from lipid-laden macrophages and thereby play an important role in the maintenance of net cholesterol balance in the arterial wall and in the reduction of pro-inflammatory responses by lipid-rich macrophages. The antiatherogenic properties of HDL have been primarily ascribed to RCT. Khera et al. recently reported that HDL efflux capacity was inversely and significantly correlated with carotid intima-media thickness (CIMT). A one-standard deviation increase in HDL efflux capacity predicted a 30% reduction in the odds for CAD. Although cholesterol efflux from macrophages represents only a small portion of total RCT, the cholesterol efflux from macrophage foam cells is probably the most relevant step with respect to preventing or reversing atherosclerosis. HDL can be separated into two major parts, i.e., pre β-(further distinguished into preβ1-, preβ2-,preβ3-HDL) and a-HDL(separated into 5 distinct subclasses HDL3c 3b 3a 2a 2b). It has been postulated that RCT indeed was the metabolic process that nascent preβ-HDL converted to mature a-HDL, following the route of preβ1-HDL→preβ2-HDL→preβ3-HDL→HDL3→HDL2[13].

The effect of HDL-C on plaque formation is complex, since HDL particles are highly heterogeneous, and exist as a spectrum of small, intermediate and large particles that differ in lipid and protein content. So the increase in plasma HDL-C does not necessarily reflect an increase in reverse cholesterol transport (RCT). Former studies from cholesteryl ester transfer protein(CETP) modulators and inhibitors such as dalcetrapib have limited efficacy to be still on the way may attributed to their concentration only on raising total HDL-C level and undesirable side effects. Results obtained in some studies, have shown that HDL quality (HDL subpopulations), rather than quantity (total HDL concentration), should be the target of future pharmacological therapies. A number of investigations have reported that, with the increase of plasma LDL-C or the decrease of plasma HDL-C concentrations or elevated TC(total cholesterol), or in some CAD patients with hyperlipidemia, or patients of CAD with diabetes, there was a general shift toward smaller-sized HDL (HDL3), which, in turn, indicates that reverse cholesterol transport might be weakened and HDL maturation might be abnormal. Significantly lower larger-sized HDL-HDL2 in CAD patients with hyperlipidemia compared with control patients, and this inverse relationship between HDL-C, HDL2, and CAD is particularly strong in men with type 2 diabetes mellitus. In type 2 diabetes patients, the difference between HDL2 in the myocardial infarction (MI) and non-MI group persists after adjustment for physical activity, alcohol intake, obesity, duration of diabetes, and glycemic control. Moreover, HDL2 deficiency has also been demonstrated to be a primary alteration in myocardial infarction patients even without other significant risk factors. The tendency that small-sized HDL3b, and HDL3a levels were significantly higher, and the large-sized HDL2a and HDL2b levels were significantly lower were also detected in ACS(acute coronary syndrome) patients. From articles on Chinese patients with elevate TC or LDL-C/HDL-C ratio, there was also a general shift toward smaller-sized HDL particles, which implied that the maturation process of HDL was blocked. Overall, accumulate evidences have demonstrated that in patients with CAD/CAD comorbid with diabetes/elevated TC levels, HDL maturation was hampered in the stage of the transformation of small-sized HDL3 to larger sized HDL2. HDL2 levels have inverse associations with the risk of acute myocardial infarction and thus to be protective factors in ischemic heart disease. It has also demonstrated that patients with high HDL2 level were better protected from atherosclerosis.

It has been demonstrate that atorvastatin 20 mg/d treatment for 8 weeks could result in a favorable modification of HDL subfraction phenotype. Treated with atorvastatin 20mg/d significantly increased the cholesterol concentration of large HDL particles and decreased the cholesterol concentration of small HDL particles although without changes of serum HDL-C level in patients with atherosclerosis. However, there are still lack of evidence on the effect of rosuvastatin treatment for HDL maturation(for the step of transformation of HDL3 to HDL2)and RCT process in CAD and Chinese patients. It has been demonstrated that Low HDL cholesterol is frequently associated with low HDL2b and high HDL cholesterol frequently associated with high HDL2b. As the investigators discussed above, compared to atorvastatin, rosuvastatin could significantly decrease LDL-C level and increase HDL-C level from baseline. So besides the basic effect of lowing LDL-C, it has a strong possibility that rosuvastatin therapy on CAD patients with hyperlipidemia could reverse the aberrant HDL maturation process via elevating lager HDL2 level, and then restore the RCT process to the normal to prevent atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with CAD undergoing quantitative coronary angiography ;
2. Patients with hyperlipidemia: TG(Triglyceride)>1.6mmol/L and/or TC(total cholesterol)>4.6mmol/L, and they didn't take antilipemic agents or steroid hormone at least three months before this trial.
3. Patients between the ages of 30 and 75 years, the functions of liver or kidney are not severe.

Exclusion Criteria:

1. Thyroid dysfunction, Liver or Biliary Tract Diseases, Acute Myocardial Infarction during the last half year, Renal Insufficiency or Kidney Failure and Cerebrovascular Trauma;
2. Drug induce Hyperlipidemia, Familial Hypercholesterolemia;
3. Having a major trauma , operation with intestines and stomach recently or the disease affecting drug absorbed;
4. Having Anaphylactic Reaction, Mental Disorders and Drinking history.
5. Taking statin, Nicotinic Acids and other drugs which can influence the level of HDL.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy endpoint is to detect the percentage change of HDL2 level by using rosuvastatin after 12 weeks in hyperlipidemia patients with CAD compared with baseline. | Visit 0 (Screening and Enrollment, 0 day);Visit 1 (4weeks);Visit 2 (8weeks);Visit 3 (12weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Xu-kai Wang, PhD, Study Chair — the Department of Cardiology, Daping Hospital, the Third Military Medical University
Locations (1):
- Xu-kai Wang, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Result] Tian L, Long S, Li C, Liu Y, Chen Y, Zeng Z, Fu M. High-density lipoprotein subclass and particle size in coronary heart disease patients with or without diabetes. Lipids Health Dis. 2012 May 15;11:54. doi: 10.1186/1476-511X-11-54. PMID 22584085
- [Result] Pirillo A, Norata GD, Catapano AL. High-density lipoprotein subfractions--what the clinicians need to know. Cardiology. 2013;124(2):116-25. doi: 10.1159/000346463. Epub 2013 Feb 20. PMID 23428644
- [Result] Navab M, Reddy ST, Van Lenten BJ, Anantharamaiah GM, Fogelman AM. The role of dysfunctional HDL in atherosclerosis. J Lipid Res. 2009 Apr;50 Suppl(Suppl):S145-9. doi: 10.1194/jlr.R800036-JLR200. Epub 2008 Oct 27. PMID 18955731
- [Result] Barter P, Gotto AM, LaRosa JC, Maroni J, Szarek M, Grundy SM, Kastelein JJ, Bittner V, Fruchart JC; Treating to New Targets Investigators. HDL cholesterol, very low levels of LDL cholesterol, and cardiovascular events. N Engl J Med. 2007 Sep 27;357(13):1301-10. doi: 10.1056/NEJMoa064278. PMID 17898099
- [Result] Katabami T, Murakami M, Kobayashi S, Matsui T, Ujihara M, Takagi S, Higa M, Ichijo T, Ohta A, Tanaka Y. Efficacy of low-dose rosuvastatin in patients with type 2 diabetes and hypo high-density lipoprotein cholesterolaemia. J Int Med Res. 2014 Apr;42(2):457-67. doi: 10.1177/0300060513507648. Epub 2014 Mar 4. PMID 24595147
- [Result] Kaneko K, Saito H, Takahashi T, Kiribayashi N, Omi K, Sasaki T, Niizeki T, Sugawara S, Akasaka M, Kubota I. Rosuvastatin improves plaque morphology in cerebral embolism patients with normal low-density lipoprotein and severe aortic arch plaque. J Stroke Cerebrovasc Dis. 2014 Jul;23(6):1682-9. doi: 10.1016/j.jstrokecerebrovasdis.2014.01.018. Epub 2014 Apr 13. PMID 24739590
- [Result] Expert Dyslipidemia Panel of the International Atherosclerosis Society Panel members. An International Atherosclerosis Society Position Paper: global recommendations for the management of dyslipidemia--full report. J Clin Lipidol. 2014 Jan-Feb;8(1):29-60. doi: 10.1016/j.jacl.2013.12.005. Epub 2013 Dec 17. PMID 24528685
- [Result] Tian L, Li C, Liu Y, Chen Y, Fu M. The value and distribution of high-density lipoprotein subclass in patients with acute coronary syndrome. PLoS One. 2014 Jan 23;9(1):e85114. doi: 10.1371/journal.pone.0085114. eCollection 2014. PMID 24465490